CLINICAL TRIAL: NCT05355064
Title: Efficacy of Oral Administration of Trehalose in Patients With Parkinson Disease in Both Idiopathic and Induced by LRRK2 Mutation
Brief Title: Efficacy of Oral Administration of Trehalose in Patients With Parkinson Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Nicola Modugno, Principal Investigator, Neuromed IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trehalose treatment in PD
Record Dates: First submitted 2021-12-18; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Trehalose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single treatment, no placebo.
  Interventions: Drug: Trehalose

INTERVENTIONS:
Drug: Trehalose — Enrolled subjects will daily take 4 g of trehalose in oral administration for 24 weeks.
  Other Names: CITOPLAS

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disease characterized by the neurodegeneration of substance nigra pars compacta (SNpc) and the formation of alpha-synuclein protein aggregates in neurons. Although most PD patients are sporadic, it is now clear that genetic factors contribute to the pathogenesis of PD. Indeed, LRRK2 G2019S mutation is one of the most common causes of familial PD. The phenotype corresponding to this mutation is a late-onset form of PD characterized by the accumulation of the N-ethylmaleimide sensitive factor (NSF) in neurons. It is due to a dysfunction of the physiological autophagy processes occurring at cellular level, mainly affecting autophagy mediated by chaperone proteins (Chaperon Mediated Autophagy, CMA), responsible for the clearance of alpha synuclein at the lysosomal level. This condition, although sensitive to treatment with L-DOPA and dopamine agonists, does not currently have any specific therapy.

Recently, in a mouse model carrying the LRRK2 mutation, it has been demonstrated that treatment with trehalose is able to reduce the accumulation of NSF deposits in neurons of various brain areas such as the substantia nigra, striatum, cortex and hippocampus. The reduction of protein aggregates correlates with intracellular molecules related to the activation of apoptotic processes in damaged neurons. Moreover, it has been found a significant improvement in motor and cognitive performance. The aim of the present study is to evaluate the safety and tolerability of trehalose in two groups of patients affected by idiopathic PD and PD carrying the LRRK2 mutation, respectively. Moreover, the investigators will collect preliminary data on the effect that this molecule potentially has on disease course in both groups. The treatment duration will be 24 weeks and the overall study duration approximately 12 months. The populations observed will be composed of subjects affected by idiopathic PD and familial PD carrying the genetically confirmed LRRK2 mutation. Enrolled subjects will daily take trehalose in oral administration. Safety will be assessed by detecting any adverse events and analyzing blood chemistry parameters. The effect of trehalose will be evaluated through periodic clinical examinations, including the administration of specific scales and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent;
* PD diagnosis according to UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (UKPDS);
* Age between 18 and 80 years (inclusive);
* Hoehn & Yahr staging > 1;

Exclusion Criteria:

* Inability to provide written informed consent;
* Diagnosis of other concomitant neurodegenerative disease;
* Concomitant treatment with drugs similar to trehalose;
* Hypersensitivity or intolerance to the active substance administered;
* Severe swallowing problems;
* Participation in other interventional studies within 30 days from the screening;
* Other medical conditions that can interfere with results or endanger the participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Clinical laboratory test results at each visit from baseline to follow-up period | 1-36 weeks
  Summary statistics for laboratory tests will be presented at baseline and at each visit. The severity of select laboratory results will be graded according the Common Terminology Criteria for Adverse Events (CTCAE).
1. Physical and neurological examination findings, at each visit. | 1-36 weeks
  Body system (General appearance, Musculo-skeletal, Cardiovascular, Lungs, Abdomen, Neurological) findings that is judged by the investigator as a clinically significant change (worsening) compared to a baseline value will be considered an adverse event coded using MedDRA

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 1-36 weeks
  To compare the efficacy of trealose therapy as measured by the sum of the MDS-UPDRS Part III score changes from Baseline to Weeks 18, 36. The score range is 0-132, where a higher score means more severe motor impairment.
Assessment of General Cognitive Functioning on the Mini Mental State Examination (MMSE) | 1- 36 weeks
  The MMSE is a 30-point questionnaire that examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. The score ranges from 0 to 30 (cut-off = 24).
The differences between the MoCa test score from baseline to follow up period | 1-36 weeks
  The MoCa test is a one page 30 points test that can be done in 10 minutes in a routine visit. The MoCa assesses several cognitive domains. The maximum score is 30.
Changes from baseline in the Quality of Life in Neurological Disorders ( NeuroQol) and EQ-5D-5L questionnaires | 1- 36 weeks
  NeuroQol will provide a means of assessing quality of life in patient populations with chronic diseases, such as PD. Europeans Quality of life questionnaire 5 dimensions ,5 levels (EQ-5D-5L) is a standardized measure of health status which provides a simple, generic measure of health for clinical and economic appraisal.

IPD SHARING:
Plan to Share IPD: No